CLINICAL TRIAL: NCT01269346
Title: A Phase 2, Multicenter, Single-Arm Study of Eribulin Mesylate With Trastuzumab as First-Line Therapy for Locally Recurrent or Metastatic Human Epidermal Growth Factor Receptor Two (HER2) Positive Breast Cancer
Brief Title: Eribulin With Trastuzumab as First-line Therapy for Locally Recurrent or Metastatic HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-208
Record Dates: First submitted 2010-12-31; First posted 2011-01-04 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Locally recurrent; metastatic HER2Positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate 1.4 mg/m2 administered as an intravenous (IV) infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle.
  Trastuzumab 8 mg/kg will be administered as in IV infusion over a 90-minute period on Day 1 of Cycle 1. Thereafter, trastuzumab 6 mg/kg will be administered as an IV infusion over a 30-minute period on Day 1 of each subsequent cycle.

SUMMARY:
This is a multicenter phase 2 study designed to evaluate the safety and efficacy of eribulin mesylate in combination with trastuzumab as first line treatment in female subjects with locally recurrent or metastatic human epidermal growth factor receptor (HER2) positive breast cancer.

ELIGIBILITY:
Key Inclusion criteria:

* Age 18 years or older
* Histologically or cytologically proven adenocarcinoma of the breast
* Subjects who have locally recurrent or metastatic disease with at least one measurable lesion
* HER2 positive as determined by score of 3 on immunohistochemistry (IHC) staining or gene amplification by fluorescence in situ hybridization (FISH).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0, 1 or 2
* At least 12 months since prior neoadjuvant or adjuvant chemotherapy
* At least 2 weeks since prior radiotherapy, endocrine therapy, trastuzumab, or lapatinib, with complete recovery from the effects of these interventions
* Adequate renal function
* Adequate bone marrow function
* Adequate liver function
* Adequate cardiac function

Key Exclusion criteria:

* Prior chemotherapy, biologic therapy, or investigational therapy for locally recurrent or metastatic HER2 breast cancer.
* Subjects who have had a prior malignancy other than carcinoma in situ of the cervix, or nonmelanoma skin cancer
* Prior exposure to greater than 360 mg/m2 doxorubicin or liposomal doxorubicin, greater than 120 mg/m2 mitoxantrone, greater than 90 mg/m2 idarubicin, or greater than 720 mg/m2 epirubicin
* Inflammatory breast cancer
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant cardiovascular impairment
* Subjects with known central nervous system (CNS) disease are not eligible, except for those subjects with treated brain metastasis.
* Subjects with metastatic disease limited to bone are ineligible unless there is at least one lytic lesion with identifiable soft tissue components that can be evaluated by computed tomography (CT) or magnetic resonance imaging (MRI)
* Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring the use of oxygen
* History of bleeding diasthesis
* Currently pregnant or breast-feeding.
* Subjects with preexisting Grade 3 or 4 neuropathy. Any peripheral neuropathy must recover to Grade less than or equal to 2 before enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Misir, Study Director — Eisai Inc.
Locations (26):
- United States (26):
  - University of Colorado, Denver, Colorado
  - Florida Cancer Care, Davie, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Peachtree Hematology Oncology Associates, PC, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Weill Cornell Breast Clinic, New York, New York
  - Raleigh Hematology Associates, Raleigh, North Carolina
  - Cancer Care of the Cascades, Bend, Oregon
  - Medical Oncology Associates of Wyoming Valley, P.C., Kingston, Pennsylvania
  - Charleston Hematology/Oncology, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - C. Michael Jones, MD, Germantown, Tennessee
  - Texas Oncology - Beaumont Marnie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology - McAllen South Second Street, McAllen, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Pensisula Cancer Institute, Newport News, Virginia
  - Columbia Basin Hematology and Oncology, Kennewick, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 participants were screened for entry into the study, of these participants 12 were screen failures and 52 were enrolled into the study and received at least one dose of study treatment.
Groups:
- Eribulin Mesylate in Combination With Trastuzumab: Eribulin Mesylate: Eribulin mesylate 1.4 mg/m^2 was administered as an intravenous (IV) infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle.
  Trastuzumab 8 mg/kg was administered as an IV infusion over a 90-minute period on Day 1 of Cycle 1. Thereafter, trastuzumab 6 mg/kg was administered as an IV infusion over a 30-minute period on Day 1 of each subsequent 21-day cycle.
Period: Treatment Phase
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Started | 52
Completed 6 Cycles | 45
Completed | 43
Not Completed | 9
Not completed — Disease progression | 3
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 2
Period: Extension Phase
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Started | 43 (Out of 52 participants randomized, only 43 continued into the Extension Phase of the study.)
Completed | 0
Not Completed | 43
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 4
Not completed — Disease progression | 22
Not completed — Physician decision or participant choice | 9
Not completed — Clinical progression | 1
Not completed — Started a prohibited con med | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least one dose of study drug.
Groups:
- Eribulin Mesylate in Combination With Trastuzumab: Eribulin Mesylate: Eribulin mesylate 1.4 mg/m^2 was administered as an intravenous (IV) infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle.
  Trastuzumab 8 mg/kg was administered as in IV infusion over a 90-minute period on Day 1 of Cycle 1. Thereafter, trastuzumab 6 mg/kg was administered as an IV infusion over a 30-minute period on Day 1 of each subsequent 21-day cycle.
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 52
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 58.7 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The Objective Response Rate (Complete Response plus Partial Response, (CR + PR)) was defined as the proportion of participants who have a best overall response of confirmed CR or PR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the Investigator. Tumor assessment was by computed tomography (CT)/magnetic resonance imaging (MRI). To assess best response (CR, PR, stable disease (SD), progressive disease (PD), or not estimable (NE)), the Investigator selected up to five measurable target lesions (2 per organ). All other lesions were identified as nontarget lesions. Each participant's overall tumor burden at Baseline was compared with subsequent measurements of the target lesions. For participants with CR or PR, changes in tumor sizes had to be confirmed by repeat evaluations performed not fewer than four weeks after the initial response assessment.
Time Frame: Baseline (within 28 days of first infusion of study drug); Treatment Phase (every 6 weeks during the first 6 cycles); Extension Phase (every 12 weeks) to PR or CR
Population: FAS included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 52
Percentage of participants | 71.2 [56.92 to 82.87]

2. Secondary Outcome: Time to First Response
Description: Time to first response was defined for participants whose best overall response was a CR or PR.
Time Frame: From date of first dose of study drug to the earliest date that CR or PR was objectively documented, assessed up to data cutoff (12 Sep 2013), up to approximately 2 years 9 months
Population: FAS included all participants who received at least one dose of study drug. Analyzed for responders (CR or PR) only.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Eribulin Mesylate in Combination With Trastuzumab: Eribulin Mesylate: Eribulin mesylate 1.4 mg/m^2 was administered as an IV infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle.
  Trastuzumab 8 mg/kg was administered as in IV infusion over a 90-minute period on Day 1 of Cycle 1. Thereafter, trastuzumab 6 mg/kg was administered as an IV infusion over a 30-minute period on Day 1 of each subsequent 21-day cycle.
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 37
Months | 1.3 [1.22 to 1.38]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined for participants whose best overall response was CR or PR. Participants who died without reported PD were considered to have progressed on the day of their death. Participants who were alive at the end of the study without reported PD were censored on the date of their last tumor assessment.
Time Frame: Date of a confirmed CR or PR was first documented to the date of PD or death (due to any cause and in the absence of PD), whichever occurred first, or date of data cutoff (12 Sep 2013), or up to approximately 2 years 9 months
Population: FAS included all participants who received at least one dose of study drug. Analyzed for responders only (n = 37).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 37
Months | 11.1 [6.70 to 17.77]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose of study drug until the date of first documentation of PD or date of death from any cause, whichever occurred first. Participants who died without reported PD were considered to have progressed on the day of their death. Participants who were lost to follow-up or alive and without reported PD at the end of study were censored on the date of their last tumor assessment.
Time Frame: Date of first dose of study drug to date of PD or death (from any cause) whichever came first, or date of data cutoff (12 Sep 2013), up to approximately 2 years 9 months
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 52
Months | 11.6 [9.13 to 13.93]

5. Secondary Outcome: Duration of Stable Disease (SD)
Description: Defined as the period from treatment start date to the date of PD or death, whichever occurred first. Participants who were alive without having PD as of the data cutoff date were censored as of their last tumor assessment. Calculated for participants who best response was SD.
Time Frame: Start of study treatment to date of PD or death, whichever occurred first, or date of data cutoff (12 Sep 2013), up to approximately 2 years 9 months
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Number analyzed (Participants) | 13
Months | 7.1 [5.55 to 13.50]

ADVERSE EVENTS:
Time Frame: From the date of signed informed consent until 30 days after discontinuation of study drug or until resolution, whichever occurred first. Up to approximately 2 years 10 months.
Description: Treatment-emergent adverse events and serious adverse events were reported. Safety Set included all participants who received at least one dose of study drug and had at least one postbaseline safety assessment. Study treatment toxicities were graded on a 5-point scale in accordance with Common Terminology Criteria for Adverse Events, version 4.0.
Arm/Group | Eribulin Mesylate in Combination With Trastuzumab
Serious Adverse Events (participants affected / at risk) | 15/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate in Combination With Trastuzumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 8
Cardiac failure chronic (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Modified radical mastectomy (Surgical and medical procedures) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate in Combination With Trastuzumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 9
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 31
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Electrocardiogram QT prolonged (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 3
Dacryostenosis acquired (Eye disorders) | 1
Dry eye (Eye disorders) | 3
Eye allergy (Eye disorders) | 2
Eye irritation (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 8
Vision blurred (Eye disorders) | 4
Visual impairment (Eye disorders) | 5
Vitreous detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 17
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Lip pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 24
Oesophagitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 9
Swollen tongue (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 4
Catheter site pain (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 8
Face oedema (General disorders) | 2
Fatigue (General disorders) | 36
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 2
Mucosal inflammation (General disorders) | 3
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 12
Pain (General disorders) | 3
Pyrexia (General disorders) | 12
Thrombosis in device (General disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Multiple allergies (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 3
Breast infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lobar pneumonia (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 7
Vulvovaginal mycotic infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Ejection fraction decreased (Investigations) | 3
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 6
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Lactose intolerance (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 3
Carpal tunnel syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 31
Paraesthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensorimotor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 9
Peroneal nerve palsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Bladder pain (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 4
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 46
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Heat rash (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Modified radical mastectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No